CLINICAL TRIAL: NCT01534624
Title: Development of Induced Pluripotent Stem Cells Carrying Monoamine Transporter Polymorphisms
Brief Title: Stem Cell Study of Genetics and Drug Addiction
Status: Completed | Type: Observational
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999912476; 12-DA-N476
Record Dates: First submitted 2012-02-15; First posted 2012-02-16 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2014-07-30

CONDITIONS: Induced Pluripotent Stem Cells
Keywords: Induced Pluripotent Stem Cell (iPS) Cell Lines; Addiction; Addiction-Associated Human Gene Variants; Dopamine Transporter
MeSH Terms: conditions — Ichthyosis prematurity syndrome; Behavior, Addictive

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

- Researchers are interested in studying the roles that genes play in drug and alcohol addiction. Genes seem to account for about half of the differences between people who become addicted to drugs and people who do not. This study will collect blood and skin cell samples. These cells will be used to develop stem cells that are useful for studying how genes are related to drug use and dependence.

Objectives:

- To study genetic and cellular differences between people who are addicted to drugs and those who are not.

Eligibility:

* Individuals between 21 and 65 years of age who do not use drugs.
* Individuals between 21 and 65 years of age who are in treatment with buprenorphine or methadone.

Design:

* Participants will be screened with a brief physical exam and medical history.
* Participants will also answer questions about physical and mental health, quality of life, and history of drug and alcohol use. A urine sample and cheek swab sample will be collected.
* Participants whose genetic samples match the study requirements will be asked to come back to provide a skin biopsy sample and a second urine sample.

DETAILED DESCRIPTION:
Background - The molecular- and cellular-based mechanisms that contribute to the initiation and development of addiction remain to be elucidated. Estimates have suggested that 40-60 percent of the vulnerability to addiction may be attributable to genetic aberrations. Multiple chromosomal regions have been linked to addiction including those containing the dopamine transporter (DAT) and vesicular monoamine transporter (VMAT2) genes. Current efforts to understand how polymorphisms in these monoamine transporters contribute to the molecular mechanisms of addiction are severely hindered by the inability to directly interrogate neural cell types from the patients. There is great potential for patient-specific iPS cell technology to profoundly impact our understanding of human development and disease by providing genetically distinct, functional sources of human cells.

Objective - The objective of the research is to develop a cell-based system whereby neural cells from afflicted individuals can be functionally assayed to interrogate the molecular mechanisms underlying addiction.

Study population Controls (non-drug users) and opioid dependent adults receiving opioid agonist therapy aged 21- 65 will be enrolled.

Design Participants demographic characteristics, psychosocial evaluation, and psychiatric, medical, and drug use histories will be characterized. DNA will be collected via cheek swabs of up to 30 potential participants for determination of dopamine transporter (DAT) and vesicular monoamine transporter (VMAT2) gene polymorphisms. Participants (N=16) with suitable polymorphisms will be asked to under go skin biopsies; 2 individuals for each of two genotypes for each gene (DAT or VMAT), i.e., 8 samples from addicts and 8 samples for control subjects. Collaborators at Case Western Reserve University will use the skin cells to derive and characterize patient-specific, induced pluripotent stem (iPS) cells that carry monoamine transporter polymorphisms for the hDAT1 and hVMAT2 genes. They will differentiate patient-specific iPS cells line into dopaminergic neurons and carry out a detailed and functional characterization of these cells to identify their molecular characteristics.

Outcome measures - Biological specimens from the addiction patients and controls will be used to derive and characterize patient-specific, induced pluripotent stem (iPS) cells that carry monoamine transporter polymorphisms. Patient-specific iPS cells lines will be differentiated into dopaminergic neurons. In follow up studies, we will characterize, compare, and functionally assay these patient-specific, iPS cell-derived dopaminergic neurons from control and addiction patients that carry polymorphisms for hDAT1 and hVMAT2 gene to investigate any possible association with dopamine neurotransmission variations and vulnerability to addiction.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. 21 to 65 years old

     Opioid dependent participant group only:
  2. enrollment in a substance abuse treatment protocol in Archway.

     Non-drug users
  3. no lifetime history of drug dependence as indicated by the screening ASI and Substance Abuse/Dependence Evaluation counselor interview.

EXCLUSION CRITERIA:

1. Relevant neurological disorders (including, but not limited to, Parkinson s disease and Huntington s disease).
2. contraindications to skin biopsy including, but not limited to, bleeding disorders, skin disorders, and immune disorders, that the MAI determines may alter the risk of the biopsy.
3. cognitive impairment severe enough to preclude informed consent or valid responses on questionnaires.
4. controls will also be excluded if they test positive for drugs or alcohol during screening or study visits.
5. unwillingness to allow samples to be kept for future research.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2012-02-07; Study Completion 2014-07-30

PRIMARY OUTCOMES:
Derive and characterize patient-specific, induced pluripotent stem (iPS) cells that carry monoamine transporter polymorphisms and differentiate them into dopaminergic neurons.

CONTACTS AND LOCATIONS:
Overall Officials: Kenzie Preston, Ph.D., Principal Investigator — National Institute on Drug Abuse (NIDA)
Locations (1):
- National Institute on Drug Abuse, Baltimore, Maryland, United States

REFERENCES:
- [Background] Hyman SE, Malenka RC. Addiction and the brain: the neurobiology of compulsion and its persistence. Nat Rev Neurosci. 2001 Oct;2(10):695-703. doi: 10.1038/35094560. PMID 11584307
- [Background] Nestler EJ. Molecular basis of long-term plasticity underlying addiction. Nat Rev Neurosci. 2001 Feb;2(2):119-28. doi: 10.1038/35053570. PMID 11252991
- [Background] Wise RA, Bozarth MA. A psychomotor stimulant theory of addiction. Psychol Rev. 1987 Oct;94(4):469-92. No abstract available. PMID 3317472